CLINICAL TRIAL: NCT00960128
Title: NordiNet® International Outcome Study-Observational Prospective Study on Patients Treated With Norditropin®
Brief Title: Observational Prospective Study on Patients Treated With Norditropin®
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GHLIQUID-3676; 2008-001674-32 (EudraCT Number)
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children; Adult Growth Hormone Deficiency; Genetic Disorder; Turner Syndrome; Foetal Growth Problem; Small for Gestational Age; Chronic Kidney Disease; Chronic Renal Insufficiency; Noonan Syndrome
MeSH Terms: conditions — Dwarfism, Pituitary; Genetic Diseases, Inborn; Turner Syndrome; Renal Insufficiency, Chronic; Noonan Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Adult cohort
  Interventions: Drug: somatropin
- B: Paediatric cohort
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — The effectiveness and safety data collection with the use of Norditropin® in daily clinical practice with adults.
  Groups: A
Drug: somatropin — The effectiveness and safety data collection with the use of Norditropin® in daily clinical practice with children.
  Groups: B

SUMMARY:
This observational study is conducted globally. The aim of the study is to investigate the effectiveness and safety of real-life treatment with Norditropin®. The study population will consist of children and adults who are on treatment with Norditropin® in accordance with normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Judged by the physician as per the Norditropin® label

Exclusion Criteria:

* Judged by the physician as per the Norditropin® label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of children and adults who are on treatment with Norditropin® in accordance with normal clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 21249 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of Norditropin® treatment on height gain (change in height) in children | Study outcomes (study endpoints) will be analysed and reported on annual basis. The mean follow up period for study outcomes is expected to be 5 years in accordance with defined duration of the study.
Effect of Norditropin® treatment on body weight and body composition in adults | Study outcomes (study endpoints) will be analysed and reported on annual basis. The mean follow up period for study outcomes is expected to be 5 years in accordance with defined duration of the study.

SECONDARY OUTCOMES:
Effect of Norditropin® treatment body weight, blood biochemistry, bone age, the endocrine system and pubertal development in children | Study outcomes (study endpoints) will be analysed and reported on annual basis. The mean follow up period for study outcomes is expected to be 5 years in accordance with defined duration of the study.
Effect of Norditropin® treatment on quality of life, blood biochemistry and the endocrine system in adults | Study outcomes (study endpoints) will be analysed and reported on annual basis. The mean follow up period for study outcomes is expected to be 5 years in accordance with defined duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (23):
- Novo Nordisk Investigational Site, Prov. de Buenos Aires, Argentina
- Novo Nordisk Investigational Site, Brussels, Belgium
- Novo Nordisk Investigational Site, Prague, Czechia
- Novo Nordisk Investigational Site, Copenhagen S, Denmark
- Novo Nordisk Investigational Site, Espoo, Finland
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Budapest, Hungary
- Novo Nordisk Investigational Site, Dublin, Ireland
- Novo Nordisk Investigational Site, Kfar Saba, Israel
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Vilnius, Lithuania
- Novo Nordisk Investigational Site, Luxembourg, Luxembourg
- Novo Nordisk Investigational Site, Alphen aan den Rijn, Netherlands
- Novo Nordisk Investigational Site, Rud, Norway
- Novo Nordisk Investigational Site, Moscow, Russia
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Malmo, Sweden
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- [Result] Weber MM, Biller BM, Pedersen BT, Pournara E, Christiansen JS, Hoybye C. The effect of growth hormone (GH) replacement on blood glucose homeostasis in adult nondiabetic patients with GH deficiency: real-life data from the NordiNet(R) International Outcome Study. Clin Endocrinol (Oxf). 2017 Feb;86(2):192-198. doi: 10.1111/cen.13256. Epub 2016 Nov 21. PMID 27736009
- [Result] Savendahl L, Pournara E, Pedersen BT, Blankenstein O. Is safety of childhood growth hormone therapy related to dose? Data from a large observational study. Eur J Endocrinol. 2016 May;174(5):681-91. doi: 10.1530/EJE-15-1017. Epub 2016 Feb 22. PMID 26903552
- [Result] Lee PA, Savendahl L, Oliver I, Tauber M, Blankenstein O, Ross J, Snajderova M, Rakov V, Pedersen BT, Christesen HT. Comparison of response to 2-years' growth hormone treatment in children with isolated growth hormone deficiency, born small for gestational age, idiopathic short stature, or multiple pituitary hormone deficiency: combined results from two large observational studies. Int J Pediatr Endocrinol. 2012 Jul 12;2012(1):22. doi: 10.1186/1687-9856-2012-22. PMID 22788856
- [Result] Hoybye C, Savendahl L, Christesen HT, Lee P, Pedersen BT, Schlumpf M, Germak J, Ross J. The NordiNet(R) International Outcome Study and NovoNet(R) ANSWER Program(R): rationale, design, and methodology of two international pharmacoepidemiological registry-based studies monitoring long-term clinical and safety outcomes of growth hormone therapy (Norditropin(R)). Clin Epidemiol. 2013 Apr 26;5:119-27. doi: 10.2147/CLEP.S42602. Print 2013. PMID 23658497
- [Result] Savendahl L, Blankenstein O, Oliver I, Christesen HT, Lee P, Pedersen BT, Rakov V, Ross J. Gender influences short-term growth hormone treatment response in children. Horm Res Paediatr. 2012;77(3):188-94. doi: 10.1159/000337570. Epub 2012 Apr 12. PMID 22508317
- [Result] Blankenstein O, Snajderova M, Blair J, Pournara E, Pedersen BT, Petit IO. Real-life GH dosing patterns in children with GHD, TS or born SGA: a report from the NordiNet(R) International Outcome Study. Eur J Endocrinol. 2017 Aug;177(2):145-155. doi: 10.1530/EJE-16-1055. Epub 2017 May 18. PMID 28522645
- [Result] Christesen HT, Pedersen BT, Pournara E, Petit IO, Juliusson PB. Short Stature: Comparison of WHO and National Growth Standards/References for Height. PLoS One. 2016 Jun 9;11(6):e0157277. doi: 10.1371/journal.pone.0157277. eCollection 2016. PMID 27280591
- [Derived] Rohrer TR, Kotnik P, Miller BS, Kelepouris N, Olsen AH, Pietropoli A, Polak M, Blair J. Better growth outcomes in GH-deficient children treated younger than 2 years of age. Endocr Connect. 2025 Sep 23;14(9):e250493. doi: 10.1530/EC-25-0493. Print 2025 Sep 1. PMID 40919719
- [Derived] Backeljauw P, Blair JC, Ferran JM, Kelepouris N, Miller BS, Pietropoli A, Polak M, Savendahl L, Verlinde F, Rohrer TR. Early GH Treatment Is Effective and Well Tolerated in Children With Turner Syndrome: NordiNet(R) IOS and Answer Program. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2653-2665. doi: 10.1210/clinem/dgad159. PMID 36947589
- [Derived] Biller BMK, Hoybye C, Carroll P, Gordon MB, Birkegard AC, Kelepouris N, Nedjatian N, Weber MM. Pregnancy outcomes in women receiving growth hormone replacement therapy enrolled in the NordiNet(R) International Outcome Study (IOS) and the American Norditropin(R) Studies: Web-Enabled Research (ANSWER) Program. Pituitary. 2021 Aug;24(4):611-621. doi: 10.1007/s11102-021-01138-3. Epub 2021 Mar 12. PMID 33709288
- [Derived] Savendahl L, Polak M, Backeljauw P, Blair JC, Miller BS, Rohrer TR, Hokken-Koelega A, Pietropoli A, Kelepouris N, Ross J. Long-Term Safety of Growth Hormone Treatment in Childhood: Two Large Observational Studies: NordiNet IOS and ANSWER. J Clin Endocrinol Metab. 2021 May 13;106(6):1728-1741. doi: 10.1210/clinem/dgab080. PMID 33571362
- [Derived] Weber MM, Gordon MB, Hoybye C, Jorgensen JOL, Puras G, Popovic-Brkic V, Molitch ME, Ostrow V, Holot N, Pietropoli A, Biller BMK. Growth hormone replacement in adults: Real-world data from two large studies in US and Europe. Growth Horm IGF Res. 2020 Feb;50:71-82. doi: 10.1016/j.ghir.2019.09.002. Epub 2019 Oct 26. PMID 31972476
- [Derived] Savendahl L, Polak M, Backeljauw P, Blair J, Miller BS, Rohrer TR, Pietropoli A, Ostrow V, Ross J. Treatment of Children With GH in the United States and Europe: Long-Term Follow-Up From NordiNet(R) IOS and ANSWER Program. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4730-4742. doi: 10.1210/jc.2019-00775. PMID 31305924
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com